CLINICAL TRIAL: NCT02086305
Title: Effects of a Transitional Palliative Care Model on Patients With End-stage Heart Failure
Brief Title: Transitional Palliative Care in End-stage Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Frances Kam Yuet WONG, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PolyU5492
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: End Stage Heart Disease; Heart Failure
Keywords: Transitional care; Supportive and palliative care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care + Transitional Care Model (Experimental): Transitional Care, Evidence-based symptom management, Protocol-driven home visit and telephone follow-up, Trained nurse case manager and volunteer partnership
  Interventions: Behavioral: Transitional Care Model; Behavioral: Usual care
- Usual Care (Active Comparator): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Transitional Care Model — Symptom assessment and management, care goal setting, post-discharge support
  Arms: Usual Care + Transitional Care Model
Behavioral: Usual care — Usual care is the routine practice in the hospital

SUMMARY:
Palliative care for end-stage organ failure patients has been included as one of the key programs to be implemented in 2011-2012 in the Hospital Authority, Hong Kong. Among all the disease groups, end-stage heart failure patients have the highest mortality rate. Patients at the end stage of heart failure have health concerns shared by other end-stage patients including cancer patients. Many guidelines, local and world-wide, have advocated a palliative approach of care for those heart failure patients who are at end stage. Studies have shown that end-stage heart failure patients tend to have frequent emergency room visits and repeated hospital admissions. Also, these patients suffer from a number of health problems that adversely affect their Quality Of Life.

There is scarcity of experimental studies informing practitioners which models work best for palliative patients in Hong Kong. There were randomized controlled trials conducted outside Hong Kong which suggest multidisciplinary approach of palliative care is possible to reduce readmissions but evidence is not present for other outcomes such as symptom control and carer burden.

In an attempt to fill knowledge gap and inform practice using evidence, this study is launched to compare the effects of a customary hospital-based palliative heart failure care and an interventional Home-based Palliative heart failure Program.

Hypothesis

* there is no difference in health care utilization for end-stage heart failure patients between the customary hospital-based group and the Home based palliative heart failure program group
* there is no difference in evaluated health outcomes (functional status, symptom intensity, and satisfaction with care) between the customary hospital-based group and the Home based palliative heart failure program group
* there is no difference in perceived health outcomes (quality of life, caregiver burden) between the customary hospital-based group and the Home based palliative heart failure program group
* there is no difference in cost effectiveness between the customary hospital-based group and the Home based palliative heart failure program group
* there is no difference In patients' lived experiences between the customary hospital-based group and the Home based palliative heart failure program group

DETAILED DESCRIPTION:
As described

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak Cantonese
* Living within the hospital service area
* Ability to be contacted by phone
* Identified as end-stage heart failure eligible for palliative care, guided by Prognostic Indicator Guidance, National Gold Standards Framework,to fulfill at least two of the indicators below:

  (i) Congestive heart failure New York Heart Association stage III or IV (ii) Patient thought to be in the last year of life by the care team (iii) Repeated hospital admissions with symptoms of heart failure (3 hospital admissions within one year) (iv) Existence of physical or psychological symptoms despite optimal tolerated therapy

Exclusion Criteria:

* Discharged to nursing home or other institution
* Inability to communicate
* Diagnosed with severe psychiatric disorders such as schizophrenia, bipolar disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization | up to 12 months
  The time from hospital discharge to hospital readmission using hospital clinical management system to retrieve data

SECONDARY OUTCOMES:
Quality of Life | baseline, 1 month, 3 months, 6 months, 12 month
  Change from baseline in quality of life on the palliative specific McGill Quality of Life Questionnaire Hong Kong version (MQOL-HK) at 1 month; change from baseline in MQOL-HK at 3 months; change from baseline in MQOL-HK at 6 months; change from baseline in MQOL-HK at 12 months
Quality of Life | Baseline, 1 month, 3 months, 6 months, 12 months
  Change from baseline in quality of life on the heart failure specific Chronic Heart Failure Questionnaire-Chinese version (CHQ) at 1 month; change from baseline in CHQ score at 3 months; change from baseline in CHQ score at 6 months; change from baseline in CHQ score at 12 months
Functional status | Baseline, 1 month, 3 months, 6 months, 12 months
  Change from baseline in functional status on the Palliative Performance Scale (PPS) at 1 month; change from baseline in PPS at 3 months; change from baseline in PPS at 6 months; change from baseline in PPS at 12 months
Symptom intensity | Baseline, 1 month, 3 month, 6 month, 12 month
  Change from baseline in symptom intensity on the Edmonton Symptom Assessment System (ESAS) at 1 month; change from baseline in ESAS score at 3 month; change from baseline in ESAS score at 6 month; change from baseline in ESAS score at 12 month.
Satisfaction with care | 1 month, 3 months, 6 months, 12 months
  Change from 1 month in satisfaction with care on the 15-item questionnaire developed by the principal investigator which validity confirmed by an expert panel and reported test-retest reliability of .87 (Sat-care) at 3 month; change from 1 month in Sat-care score at 6 months; change from 1 month in Sat-care score at 12 months
Caregiver burden | Baseline, 1 month, 3 months, 6 months, 12 months
  Change from baseline in caregiver burden on the Zarit Caregiver Burden Scale (ZCBS) at 1 month; change from baseline in ZCBS score at 3 months; change from baseline in ZCBS score at 6 months; change from baseline in ZCBS score at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frances KY Wong, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- Hong Kong (3):
  - Grantham Hospital, Hong Kong
  - Haven Of Hope Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

REFERENCES:
- [Derived] Wong FKY, So C, Ng AYM, Lam PT, Ng JSC, Ng NHY, Chau J, Sham MMK. Cost-effectiveness of a transitional home-based palliative care program for patients with end-stage heart failure. Palliat Med. 2018 Feb;32(2):476-484. doi: 10.1177/0269216317706450. Epub 2017 Apr 24. PMID 28434275
- [Derived] Ng AY, Wong FK, Lee PH. Effects of a transitional palliative care model on patients with end-stage heart failure: study protocol for a randomized controlled trial. Trials. 2016 Mar 31;17:173. doi: 10.1186/s13063-016-1303-7. PMID 27037096